CLINICAL TRIAL: NCT01595789
Title: Adding Liraglutide to the Backbone Therapy of Biguanide in Patients With Coronary Artery Disease and Newly Diagnosed Type-2 Diabetes
Brief Title: The Effect of Liraglutide on the Treatment of Coronary Artery Disease and Type 2 Diabetes
Acronym: AddHope2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Haugaard, Steen Bendix, M.D., DMSc (Individual)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BBHAH-2011430; 2011-005405-78 (EudraCT Number)
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease; Diabetes Mellitus, Type 2
Keywords: Coronary Artery Disease; Diabetes Mellitus; Left ventricular ejection fraction; Beta-cell function
MeSH Terms: conditions — Coronary Artery Disease; Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo + metformin (Placebo Comparator)
  Interventions: Drug: Placebo
- Liraglutide + metformin (Active Comparator)
  Interventions: Drug: Liraglutide

INTERVENTIONS:
Drug: Liraglutide — Liraglutide injection pen is administered by the participant once daily by subcutaneous injection. It is given independent of meals. The starting dose is 0.6 mg. After 2 weeks the dose will be increased to 1.2 mg. The dose will be further increased after 4 weeks to 1.8 mg. After a total of 12 weeks of treatment, a wash-out period of 2 weeks follows. Subsequently, the participant will be crossed over to a second period of 12 weeks of treatment with placebo.
  Other Names: Brand name: Victoza; Active substance: liraglutide; EMA Product number: EMEA/H/C/001026; ATC Code: A10BX07
  Arms: Liraglutide + metformin
Drug: Placebo — Volume-matched placebo injection pen is administered by the participant once daily by subcutaneous injection. It is given independent of meals. The starting dose is 0.6 mg volume-matched placebo. After 2 weeks the dose will be increased to 1.2 mg. The dose will be further increased after 4 weeks to 1.8 mg. After a total of 12 weeks of treatment, a wash-out period of 2 weeks follows. Subsequently, the participant will be crossed over to a second period of 12 weeks of treatment with liraglutide.
  Arms: Placebo + metformin

SUMMARY:
The purpose of this study is to investigate the effect of combined glucagon-like-peptide-1 (GLP-1) analogue and metformin therapy on glucose metabolic and cardiovascular endpoints compared to metformin monotherapy in patients with coronary artery disease (CAD) and newly diagnosed type 2 diabetes (T2D).

It is hypothesized that GLP-1 analogue added to backbone therapy of metformin in CAD patients with T2D will improve beta-cell function, left ventricular ejection fraction (LVEF), heart rate variability and lower 24h blood pressure among other selected endpoints.

The present study on CAD patients with newly diagnosed T2D will address these selected endpoints during an investigator initiated, randomized, double blind, crossover, placebo-controlled 12 + 12 weeks intervention study with a 2 week wash-out period.

DETAILED DESCRIPTION:
The total study period for each patient will be 26 weeks (12 plus 12 weeks of intervention with a 2 week wash-out period).

The endpoints will be evaluated at baseline (week 0), at week 12, at week 14 (following 2 weeks of wash-out) and finally at week 26.

ELIGIBILITY:
Inclusion Criteria:

1. Stable CAD documented by one of the following:

   * Previous MI (a minimum of 6 weeks after an acute MI)
   * Previous coronary revascularization
   * CAD confirmed by an abnormal coronary angiography (CAG) or CT-angiography showing stenosis > 50% of any major coronary arteries.
2. Body mass index (BMI) >/= 25,0 kg/m2
3. Age >/= 18 years and </= 85 years
4. Type 2 diabetes diagnosed by one of the following criteria:

   * HbA1c >/= 6.5%
   * HbA1c < 6.5 % and fasting plasma glucose >/= 7.0 mmol/l (confirmed)
   * HbA1c < 6.5 % and a 2 h plasma glucose value during OGTT >/= 11.1 mmol/l

The data for glucose metabolism are accepted provided that they have been obtained within 24 months prior to inclusion of the patient. The glucose metabolic categories are defined by ADA and WHO criteria.

Exclusion Criteria:

* Type 1 diabetes mellitus defined as C-peptide < 450 pM
* Previously diagnosed diabetes mellitus for more than 24 months prior to the screening procedure for this trial, except from gestational diabetes
* Use of more than 2 types of oral antidiabetic medication and/or use of parenteral antidiabetic medication in the period of 3 months prior to the screening visit. It is accepted that the patient continues his usual antidiabetic medication after the screening visit but antidiabetic medication must be discontinued 2 weeks prior to the baseline visit.
* Significant heart disease (NYHA > 2; Ejection Fraction < 40% and unstable angina pectoris) and known severe valve disease
* Documented atrial fibrillation or atrial flutter within 6 weeks previous to the screening. Paroxysmal atrial fibrillation is accepted if sinus rhythm is achieved at the screening.
* Uncontrolled arterial hypertension (> 180/100 mmHg) at the time of screening
* Liver (transaminases greater than x 2 the upper normal level) or renal diseases (eGFR < 60 ml/min)
* Amylase greater than x 3 the upper reference value
* Any chronic medical condition to unduly increase risk for the potential enrollee as judged by study investigators
* Dysregulated myxedema or hyperthyroid condition defined by a value of TSH < 0,1 and > 10,0 milli U/L
* Anemia (< 85% of lower normal limit), leucopenia (< 85% of lower normal limit), or thrombocytopenia (< 85% of lower normal limit)
* Pregnancy or failure to comply with contraception planning within two years, or breastfeeding
* Abuse of alcohol or drugs, or any other co-existing condition that would make patients unsuitable to participate in the study, as judged by the investigators
* Use of immunosuppressive therapy in the preceding 12 months
* Chronic pancreatitis or previous acute pancreatitis
* Known or suspected hypersensitivity to trial product(s) or related products
* Treatment with oral glucocorticoids, calcineurin inhibitors, or dipeptidyl peptidase 4 (DPP4) inhibitors, or other GLP-1 mimetics (e.g. exenatide), which in the Investigator's opinion could interfere with glucose metabolism
* Cancer (except basal cell skin cancer or squamous cell skin cancer) or any other clinically significant disorder, which in the Investigator's opinion could interfere with the results of the trail
* Inflammatory bowel disease
* Previous bowel resection
* Clinical signs of diabetic gastroparesis
* Plasma calcium-ion >/= 1,45 mmol/L
* Plasma calcitonin >/= 50 ng/L
* Subjects with personal or family history of medullary thyroid carcinoma or a personal history of multiple endocrine neoplasia type 2
* Refusal to sign informed consent.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2012-05; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Beta-cell function | after 12 weeks of intervention
  Beta-cell function (disposition index) as measured during an intravenous glucose tolerance test (By Bergman Minimal Model)
LVEF | after 12 weeks of intervention
  Changes in LVEF assessed by dobutamine stress echocardiography

SECONDARY OUTCOMES:
Glucagon, incretin, glucose, NEFA, insulin and C-peptide response during meal test | Baseline (week 0), week 12, week 14, week 26
Insulin sensitivity (Si), acute insulin and C-peptide response to intravenous glucose (AIRg, ACRg), glucose clearance (Kg), glucose effectiveness (Sg) and hepatic extraction of insulin (HEXi) | Baseline (week 0), week 12, week 14, week 26
  Insulin sensitivity (Si), acute insulin and C-peptide response to intravenous glucose (AIRg, ACRg), glucose clearance (Kg), glucose effectiveness (Sg) and hepatic extraction of insulin (HEXi) derived from a standard frequent sampling intravenous glucose tolerance test (FSIGT, Minimal model)
CRP, TNF-alfa and IL-6 in plasma and gene expression of IL6 and TNF-alfa in subcutaneous fat | Baseline (week 0), week 12, week 14, week 26
Non esterified fatty acids (NEFA) | Baseline (week 0), week 12, week 14, week 26
  NEFA during FSIGT by use of NEFA minimal model
Heart rate variability (HRV) | Baseline (week 0), week 12, week 14, week 26
  HRV i.e. SDNN (standard deviation of all normal RR interval) assessed during HOLTER monitoring
Maximal velocity of the myocardium in systole (s´) and in diastole (e´) | Baseline (week 0), week 12, week 14, week 26
  Maximal velocity of the myocardium in systole (s´) and in diastole (e´) during the dobutamine stress test
Changes in exercise tolerance test variables: Total exercise duration (sec), time to limiting angina (sec) and time to 1 mm ST-segment depression (sec) | Baseline (week 0), week 12, week 14, week 26
  Changes in exercise tolerance test variables: Total exercise duration (sec), time to limiting angina (sec) and time to 1 mm ST-segment depression (sec)
ST-depression and ectopic activity | Baseline (week 0), week 12, week 14, week 26
  ST-depression and ectopic activity assessed during 24h HOLTER monitoring
Diurnal blood pressure | Baseline (week 0), week 12, week 14, week 26
Diastolic heart function (E/E*) | Baseline (week 0), week 12, week 14, week 26
  Diastolic heart function (E/E*) in rest and during stress

CONTACTS AND LOCATIONS:
Overall Officials: Steen B Haugaard, M.D., DMSc, Study Director — Amager Hospital; Ahmad Sajadieh, M.D., DMSc, Principal Investigator — University Hospital Bispebjerg and Frederiksberg
Locations (1):
- Copenhagen University Hospital, Bispebjerg, Copenhagen, Bispebjerg, Denmark

REFERENCES:
- [Derived] Kumarathurai P, Sajadieh A, Anholm C, Kristiansen OP, Haugaard SB, Nielsen OW. Effects of liraglutide on diastolic function parameters in patients with type 2 diabetes and coronary artery disease: a randomized crossover study. Cardiovasc Diabetol. 2021 Jan 7;20(1):12. doi: 10.1186/s12933-020-01205-2. PMID 33413428
- [Derived] Anholm C, Kumarathurai P, Jurs A, Pedersen LR, Nielsen OW, Kristiansen OP, Fenger M, Holst JJ, Madsbad S, Sajadieh A, Haugaard SB. Liraglutide improves the beta-cell function without increasing insulin secretion during a mixed meal in patients, who exhibit well-controlled type 2 diabetes and coronary artery disease. Diabetol Metab Syndr. 2019 May 31;11:42. doi: 10.1186/s13098-019-0438-6. eCollection 2019. PMID 31164926
- [Derived] Kumarathurai P, Anholm C, Fabricius-Bjerre A, Nielsen OW, Kristiansen O, Madsbad S, Haugaard SB, Sajadieh A. Effects of the glucagon-like peptide-1 receptor agonist liraglutide on 24-h ambulatory blood pressure in patients with type 2 diabetes and stable coronary artery disease: a randomized, double-blind, placebo-controlled, crossover study. J Hypertens. 2017 May;35(5):1070-1078. doi: 10.1097/HJH.0000000000001275. PMID 28129251
- [Derived] Kumarathurai P, Anholm C, Larsen BS, Olsen RH, Madsbad S, Kristiansen O, Nielsen OW, Haugaard SB, Sajadieh A. Effects of Liraglutide on Heart Rate and Heart Rate Variability: A Randomized, Double-Blind, Placebo-Controlled Crossover Study. Diabetes Care. 2017 Jan;40(1):117-124. doi: 10.2337/dc16-1580. Epub 2016 Oct 19. PMID 27797930
- [Derived] Kumarathurai P, Anholm C, Nielsen OW, Kristiansen OP, Molvig J, Madsbad S, Haugaard SB, Sajadieh A. Effects of the glucagon-like peptide-1 receptor agonist liraglutide on systolic function in patients with coronary artery disease and type 2 diabetes: a randomized double-blind placebo-controlled crossover study. Cardiovasc Diabetol. 2016 Jul 26;15(1):105. doi: 10.1186/s12933-016-0425-2. PMID 27455835
- [Derived] Anholm C, Kumarathurai P, Klit MS, Kristiansen OP, Nielsen OW, Ladelund S, Madsbad S, Sajadieh A, Haugaard SB; AddHope2 Trial Study Group. Adding liraglutide to the backbone therapy of biguanide in patients with coronary artery disease and newly diagnosed type-2 diabetes (the AddHope2 study): a randomised controlled study protocol. BMJ Open. 2014 Jul 16;4(7):e005942. doi: 10.1136/bmjopen-2014-005942. PMID 25031198